CLINICAL TRIAL: NCT06404021
Title: Randomized Open-label Single-center Trial on Remote Assistance Implementing Certified Specialized Engineers During Interventional Cardiology Procedures
Brief Title: Electronic Device Implantation Through Remote Guidance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calabria (Other)
Responsible Party: Principal Investigator, Antonio Curcio, MD, PhD, University of Calabria
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: #224
Record Dates: First submitted 2024-04-26; First posted 2024-05-08 (Actual); Results first posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Telemedicine; Heart Failure; Defibrillators
Keywords: electrophysiology; remote monitoring; technical support; device
MeSH Terms: conditions — Heart Failure | interventions — Engineering

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional cardiology procedures with engineer in remote support (Experimental)
  Interventions: Other: interventional cardiology procedures with proctoring system
- Interventional cardiology procedures with engineer in the electrophysiology laboratory (Active Comparator)
  Interventions: Other: interventional cardiology procedures with engineer in the electrophysiology laboratory

INTERVENTIONS:
Other: interventional cardiology procedures with proctoring system — Interventional procedures are performed by utilizing a monitoring platform that provides real-time support without engineer in the electrophysiology laboratory
  Arms: Interventional cardiology procedures with engineer in remote support
Other: interventional cardiology procedures with engineer in the electrophysiology laboratory — Biomedical engineers supervise the performance of interventional cardiology procedures in the electrophysiology laboratory.
  Arms: Interventional cardiology procedures with engineer in the electrophysiology laboratory

SUMMARY:
Implantable cardioverter defibrillators (ICD) and cardiac resynchronization therapy defibrillator (CRT-D) implants are limited by availability and costs of field clinical specialist (FCS) bioengineers. This study explores feasibility of remotely supported implantations through an internet based platform, aiming at enhancing efficiency and overcoming geographical or pandemic related barriers. The first phase of the study included programming and phantom assessments in 20 cases followed by 10 remote guided CRT-D and ICD implantations in additional heart failure patients, compared to 20 procedures with FCS on site. Data analysis revealed no significant differences in acute outcomes or electronic parameters at one year follow-up compared to on-site FCS. Finally, this study demonstrates the safety after testing at one year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Patients under 85 years
* Patients already implanted with defibrillator and admitted to cardiology division for others invasive procedures
* Patients undergoing defibrillator or cardiac resynchronization therapy defibrillator implantation
* Patients who signed written informed consent

Exclusion Criteria:

* Pacemaker dependent patients
* Patients who underwent generator replacement procedures

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Curcio, Principal Investigator — University of Calabria
Locations (1):
- "Magna Graecia" University of Catanzaro, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Interventional Cardiology Procedures With Engineer in Remote Support | Interventional Cardiology Procedures With Engineer in the Electrophysiology Laboratory
Started | 10 | 20
Completed | 10 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: both genders and in range 18 ÷ 85 years of age
Groups:
- Total: Total of all reporting groups
Arm/Group | Interventional Cardiology Procedures With Engineer in Remote Support | Interventional Cardiology Procedures With Engineer in the Electrophysiology Laboratory | Total
Number analyzed (Participants) | 10 | 20 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 20 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (11) | 64 (11) | 64 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 7 | 14 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 20 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 10 | 20 | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Interventional Procedures Successfully Completed
Description: Investigators are going demonstrate the feasibility of cardiology interventional procedures using a proctoring system, comparing them to on site operations carried out by a biomedical engineer. For this purpose engineers develop a system for remote technical support with dedicated computer room, multimedia information system and multi angles cameras, located at the boarders of the electrophysiology lab. In the preclinical step phantom are used for approaching all types of materials and equipment that are going to be used in interventional procedures. Each procedure is considered complete and feasible when the measurements of the electronic parameters of all implanted leads are optimal, in particular, when the pacing function was effective (pacing threshold less than 1 Volt @ 0.5 millisecond).
Time Frame: From enrollment to the end of treatment at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional Cardiology Procedures With Engineer in Remote Support | Interventional Cardiology Procedures With Engineer in the Electrophysiology Laboratory
Number analyzed (Participants) | 10 | 20
Participants | 10 | 20

2. Primary Outcome: Mean Pacing Threshold at 12-Month Follow-Up
Description: The outcome assesses the mean pacing threshold at 12-month follow-up, used as an indicator of long-term electrical stability of implanted cardiac leads. Stable pacing thresholds suggest proper lead function and adequate myocardial contact over time.
Time Frame: 12-month follow-up visit
Measure: Mean (Standard Deviation); unit: Volt
Arm/Group | Interventional Cardiology Procedures With Engineer in Remote Support | Interventional Cardiology Procedures With Engineer in the Electrophysiology Laboratory
Number analyzed (Participants) | 10 | 20
Volt | 0.42 (0.12) | 0.42 (0.098)

3. Primary Outcome: Fluoroscopy Time (Minutes) During Cardiac Device Implantation With or Without Remote Assistance
Description: Fluoroscopy time (FT), expressed in minutes, is used as a surrogate measure of procedural efficiency and radiation exposure. The FT corresponds to the skin-to-skin time and is recorded from the beginning of X-ray emission to the end of the cardiac device implantation procedure. Data are compared between two groups: procedures performed with onsite presence of the biomedical engineer and those executed with remote technical assistance through the telemedicine support system.
Time Frame: During the interventional procedure up to 2 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Interventional Cardiology Procedures With Engineer in Remote Support | Interventional Cardiology Procedures With Engineer in the Electrophysiology Laboratory
Number analyzed (Participants) | 10 | 20
minutes | 6 (4) | 8 (8)

4. Primary Outcome: Electrophysiology Laboratory Occupancy
Description: Investigators determined the duration of interventional procedures in minutes and compared this result both for standard and telemedicine driven approach.
Time Frame: The time in minutes during procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Interventional Cardiology Procedures With Engineer in Remote Support | Interventional Cardiology Procedures With Engineer in the Electrophysiology Laboratory
Number analyzed (Participants) | 10 | 20
minutes | 84 (6.5) | 103 (28)

ADVERSE EVENTS:
Time Frame: From device implantation through 12 months post-procedure, assessed at baseline, 6 months, and 12 months
Description: All patients could be at risk of adverse events. All participants were monitored for serious adverse events throughout the study period.
Arm/Group | Interventional Cardiology Procedures With Engineer in Remote Support | Interventional Cardiology Procedures With Engineer in the Electrophysiology Laboratory
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/20
Other Adverse Events (participants affected / at risk) | 0/10 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/21/NCT06404021/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/21/NCT06404021/ICF_001.pdf